CLINICAL TRIAL: NCT05387681
Title: An Exploratory Clinical Study of Short-course Radiotherapy Combined With Envafolimab, Endostatin and SOX Regimen for Neoadjuvant Treatment of Resectable Locally Advanced Gastric/Gastroesophageal Junction Adenocarcinoma
Brief Title: Preoperative Short Course Radiotherapy With Envafolimab, Endostatin and SOX Regimen in Locally Advanced Gastric
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Tao Zhang, Chief of Cancer Center, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SMA-GC-003V
Record Dates: First submitted 2022-05-12; First posted 2022-05-24 (Actual); Last update posted 2022-05-24 (Actual); Status verified 2022-05

CONDITIONS: Gastric/Gastroesophageal Junction Adenocarcinoma; Radiotherapy; Immunotherapy
Keywords: neoadjuvant，gastric
MeSH Terms: interventions — envafolimab; Endostatins

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Envafolimab, Endostatin and SOX regimen (Experimental): Preoperative short course radiotherapy with Envafolimab, Endostatin and SOX regimen
  Interventions: Drug: Envafolimab

INTERVENTIONS:
Drug: Envafolimab — short course radiotherapy ：5*5Gy (25Gy/5F) ； Envafolimab：300 mg, subcutaneously, D1, Q3W; Endostatin ：210mg (14 doses), CIV continuously pumped for 72h, Q3W; chemotherapy：SOX regimen
  Other Names: Endostatin

SUMMARY:
This is a single-arm, exploratory clinical study to evaluate the efficacy and safety of Preoperative short course radiotherapy with Envafolimab, Endostatin and SOX regimen in resectable locally advanced gastric/gastroesophageal junction adenocarcinoma.

DETAILED DESCRIPTION:
All eligible subjects will receive 5*5Gy (25Gy/5F) fractionated radiotherapy, rest for 1 week, 3 cycles of Envafolimab, Endostatin and SOX regimen, and radical surgery 2 to 4 weeks after completion of the last neoadjuvant therapy, according to the study plan. Each patient will be followed up 12 months after initiation of treatment in the study. Whether the subjects need adjuvant therapy after surgery and the adjuvant treatment plan are determined by the investigator. All subjects were required to complete the study follow-up plan after surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Signed written informed consent before enrollment; 2.18 years old ≤75 years old, male or female; 3. Initially diagnosed locally advanced gastric/gastroesophageal junction adenocarcinoma confirmed by tissue or pathology; 4. Without systemic treatment; 5. Patients diagnosed as CT2-4an + M0 according to endoscopic ultrasonography or enhanced CT/MRI scan cTNM were assessed by researchers as suitable for neoadjuvant therapy + radical surgery. AJCC/UICC Version 8 was used for TNM pathological staging (pTNM).

6.ECOG PS score: 0 ~ 1; 7. The expected survival time is more than 6 months; 8. The function of vital organs meets the following requirements (excluding any blood components and cell growth factors within 14 days) :

1. Blood routine:

   Neutrophils ≥1.5×109/L Platelet count ≥100×109/L Hemoglobin ≥ 90g/L;
2. Liver and kidney function:

Serum creatinine (SCr) ≤ 1.5 times the upper limit of normal value (ULN) or creatinine clearance ≥50 mL /min (Cockcroft-Gault formula); Total bilirubin (TBIL) ≤ 1.5 times normal upper limit (ULN); Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) levels ≤ 2.5 times the upper limit of normal value (ULN) (≤5ULN if abnormal liver function is due to liver metastasis); Urine protein & lt; 2 +; If urine protein ≥2+, 24-hour urine protein quantification must be ≤1g; 9. Normal coagulation function, no active bleeding and thrombotic diseases

1. International standardized ratio INR≤1.5×ULN;
2. Partial thrombin time APTT≤1.5×ULN;
3. Prothrombin time PT≤1.5×ULN; 10. Women of non-surgical sterilization or childbearing age are required to use a medically approved contraceptive method (such as an intrauterine device, birth control pill or condom) during the study period and for three months after the study period; The serum or urine HCG test of female patients of reproductive age who were not undergoing surgical sterilization must be negative within 7 days prior to study enrollment. And must be non lactation period; Male patients of non-surgical sterilization or reproductive age are required to consent with their spouse to use a medically approved contraceptive method during the study treatment period and for 3 months after the study treatment period 11. The subjects voluntarily participated in the study with good compliance and follow-up for safety and survival.

Exclusion Criteria:

1. The subject has previous or co-existing malignancies (except cured basal cell carcinoma of the skin and carcinoma in situ of the cervix);
2. Previous treatment with other PD-1/PD-L1 inhibitors could not be included; Subject is known to have a prior allergy to large protein preparations, or is known to be allergic to the drug ingredient used;
3. The subjects exist any active autoimmune disease or a history of autoimmune disease (such as the following, but not limited to: autoimmune hepatitis, interstitial pneumonia, uveitis, enteritis, hepatitis, the pituitary gland inflammation, vasculitis, nephritis, thyroid function hyperfunction, thyroid function is reduced, always had thyroid surgery must be incorporated into; Subjects with vitiligo or asthma in complete remission during childhood without any intervention as adults could be included; Subjects with asthma requiring medical intervention with bronchodilators were excluded);
4. Subject is receiving immunosuppressant, or systemic, or absorbable local hormone therapy for immunosuppression purposes (dose > 10mg/ day of prednisone or other equivalent hormone) and continued to use within 2 weeks prior to enrollment;
5. Clinical ascites or pleural effusion requiring therapeutic puncture or drainage;
6. Patients with cardiac clinical symptoms or diseases that are not well controlled, such as :(1) nyha class 2 or more heart failure (2) unstable angina pectoris (3) myocardial infarction within 1 year (4) clinically significant ventricular or ventricular arrhythmias requiring treatment or intervention;
7. Within 14 days before the first administration of the study drug, Chinese herbal medicines or proprietary Chinese medicines approved by the National Medical Products Administration of China (NMPA) with antitumor activity, regardless of cancer type;
8. Subject has active infection or unexplained fever during screening but prior to initial administration & GT; 38.5 degrees (the investigator judged that the fever caused by the tumor could be included in the study);
9. Patients with past or present objective evidence of pulmonary fibrosis, interstitial pneumonia, pneumoconiosis, radioactive pneumonia, drug-associated pneumonia, known active tuberculosis, severely impaired lung function, etc.;
10. Subjects with congenital or acquired immune deficiency (such as HIV infection, HIV 1/2 antibody positive);
11. Patients with acute or chronic active Hepatitis B (HBsAg or core antibody.HBcAb) should be tested for Hepatitis B virus (HBV)DNA, such as HBV DNA copy number ≤2×103 copy number/mL or ≤200 IU/ mL or lower than the detection limit can be included. HBsAg (+) subjects should receive anti-HBV therapy throughout study drug therapy to avoid viral activation. Subjects who are resistant to HBc(+), HBsAg(-), anti-HBS (-), and HBV viral load (-) do not need prophylactic anti-HBV therapy, but should be closely monitored for virus reactivation;
12. Acute or chronic active Hepatitis C Virus (HCV), that is, HCV antibody positive and HCV RNA levels above the detection limit;
13. Received live vaccine less than 4 weeks prior to study administration or possibly during the study period;
14. The subject has a known history of psychotropic drug abuse, alcoholism or drug abuse;
15. Known Her2 positive;
16. Prone to stomach bleeding; Patients with any evidence or history of bleeding; Patients with any bleeding or bleeding event ≥CTCAE grade 3 within 4 weeks prior to grouping had unhealed wounds, ulcers or fractures;
17. Researchers think that should be left out in this study, the researchers determine, for example, the subjects have other factors that may result in this study were forced to midway termination, such as, other serious disease (including mental illness) need to merge treatment, there are serious abnormal laboratory examination, accompanied by factors such as family or society, will affect the safety of the subjects, or information and the collection of the sample.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2022-05-30 (Estimated); Primary Completion 2023-07-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
pathological complete response (pCR) | one year
  Pathological complete response (pCR) is defined as the absence of residual invasive cancer on hematoxylin and eosin evaluation of the complete resected breast specimen and all sampled regional lymph nodes following completion of neoadjuvant systemic therapy (i.e., ypT0/Tis ypN0 in the current AJCC staging system)

SECONDARY OUTCOMES:
R0 resection rates | one year
  R0 resection was performed if there was no visible tumor residue within 1 mm of the surgical margin.
pathological partial response(MPR) | one year
  It was defined as ≤ 10% remaining viable tumor cells at surgical resection of the primary tumor

CONTACTS AND LOCATIONS:
Overall Officials: Tao Zhang, MD, Principal Investigator — Cancer Center, Union Hospital, Tongji Medical College

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Li J, Deng Y, Zhang W, Zhou AP, Guo W, Yang J, Yuan Y, Zhu L, Qin S, Xiang S, Lu H, Gong J, Xu T, Liu D, Shen L. Subcutaneous envafolimab monotherapy in patients with advanced defective mismatch repair/microsatellite instability high solid tumors. J Hematol Oncol. 2021 Jun 21;14(1):95. doi: 10.1186/s13045-021-01095-1. PMID 34154614